CLINICAL TRIAL: NCT03412539
Title: Mechanism of Effectiveness of Neurosurgery Treatments for Durable Pain
Status: Available | Type: Expanded Access
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, michal roll, Dr Ido Strauss Neurosurgeon, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-0354-17-TLV
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Oncology Problem
Keywords: resistant pain

STUDY DESIGN:
Expanded Access Types: Individual

SUMMARY:
The participants in the study are patients who undergo surgery to damaged nerve transmission and processing system in the nervous system as part of the routine clinical treatment that will not be affected by the proposed study. Patients who are candidates for procedures are referred from all over the country and undergo a multidisciplinary evaluation in the framework of the Palliative Pain Management Clinic, which operates exclusively in Israel at the Sourasky Medical Center in Tel Aviv.

DETAILED DESCRIPTION:
The participants in the study are patients who undergo surgery to damaged nerve transmission and processing system in the nervous system as part of the routine clinical treatment that will not be affected by the proposed study. Patients who are candidates for procedures are referred from all over the country and undergo a multidisciplinary evaluation in the framework of the Palliative Pain Management Clinic, which operates exclusively in Israel at the Sourasky Medical Center in Tel Aviv.

During the preoperative evaluation, patients will be given an explanation about the possibility of participating in the study. Patients who agree to participate will sign an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing neurosurgical surgery for resistant pain
* Ability to sign informed consent form for participation in the study
* A functional level is sufficient for cooperation and the performance of various tasks before and after surgery, including performing MRI's, answering pain questioners, and neuropsychological evaluations.

Exclusion Criteria:

* Refusal to participate
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery, Tel-Aviv Sourasky MC, Tel Aviv, Israel